CLINICAL TRIAL: NCT04777643
Title: Sex Differences in Neural Response to Cannabidiol
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2000029579
Record Dates: First submitted 2021-02-25; First posted 2021-03-02 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: CBD; Neural Responses
MeSH Terms: interventions — Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cannabidiol (Experimental): Participants will receive a single 600mg oral dose of Epidiolex (cannabidiol) 2 hours prior to fMRI scanning.
  Interventions: Drug: Cannabidiol
- Placebo (Placebo Comparator): Participants will receive a single oral dose of placebo 2 hours prior to fMRI scanning.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Cannabidiol — Participants will receive a single 600mg oral dose of Epidiolex (cannabidiol) 2 hours prior to fMRI scanning.
  Arms: Cannabidiol
Other: Placebo — Participants will receive a single oral dose of placebo 2 hours prior to fMRI scanning.
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, within-subjects, cross-over design to assess neural changes following a single dose of cannabidiol (CBD) (600mg) versus placebo among healthy female volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Female, aged 18-65
4. In good general health as evidenced by medical history and medically eligible to receive CBD, as determined by the licensed physician, Dr. Ayana Jordan
5. Body Mass Index between 18.5 and 30
6. For females of reproductive potential: agreement to use highly effective contraception during study participation and/or negative pregnancy test prior to fMRI scanning

Exclusion Criteria:

1. Recent use of cannabis (any past month use)
2. Lifetime history of cannabis use disorder
3. Lifetime history of chronic pain disorder
4. Current DSM-5 disorder, as determined via Structured Clinical Interview (SCID-5)
5. Presence of any contraindication to MRI scanning
6. Known allergic reactions to cannabidiol
7. Lifetime use of Epidiolex
8. Currently taking any medications that could interact with cannabidiol
9. Current smoker or tobacco use >1x/week
10. Not fluent in English
11. Less than 6th grade reading level

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Females only
Enrollment: 19 (Actual)
Dates: Start 2022-06-07 (Actual); Primary Completion 2023-04-27 (Actual); Study Completion 2023-04-27 (Actual)

PRIMARY OUTCOMES:
Amygdala activation during stress | fMRI will begin 2 hours post-drug administration and will last no more than 1 hour.
  Participants will complete 1 fMRI scan following CBD administration and another fMRI scan following placebo administration. During each scan, participants will complete the Emotion Regulation Task (ERT). The first primary outcome measure will be amygdala response during the negative emotionality contrast of the ERT during their CBD relative to their placebo scan.
Insula activation during social exclusion | fMRI will begin 2 hours post-drug administration and will last no more than 1 hour.
  Participants will complete 1 fMRI scan following CBD administration and another fMRI scan following placebo administration. During each scan, participants will complete the Cyberball Task. The second primary outcome measure will be insula response during the exclusion versus inclusion contrast of the Cyberball Task during their CBD relative to their placebo scan.

SECONDARY OUTCOMES:
Patterns of amygdala functional connectivity during stress | fMRI will begin 2 hours post-drug administration and will last no more than 1 hour.
  Participants will complete 1 fMRI scan following CBD administration and another fMRI scan following placebo administration. During each scan, participants will complete the Emotion Regulation Task (ERT). The first secondary outcome measure will be participants' pattern of seed-based functional connectivity with the amygdala during the negative emotionality contrast of the ERT during their CBD relative to their placebo scan.
Patterns of insula functional connectivity during social exclusion | fMRI will begin 2 hours post-drug administration and will last no more than 1 hour.
  Participants will complete 1 fMRI scan following CBD administration and another fMRI scan following placebo administration. During each scan, participants will complete the Cyberball Task. The second secondary outcome measure will be participants' pattern of seed-based functional connectivity with the insula during the exclusion versus inclusion contrast of the Cyberball Task during their CBD relative to their placebo scan.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah D. Lichenstein, PhD, Principal Investigator — Yale University
Locations (1):
- Yale School of Medicine, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Because this is a pilot project, we do not plan to share to data. Pending the results of the pilot project, we hope to pursue funding for a larger study to examine sex differences in neural response to CBD more directly (including both male and female participants) and on a larger scale (larger sample than pilot project), and we will plan to make these data available to other researchers.